CLINICAL TRIAL: NCT02400580
Title: Intravenous Acetaminophen Versus Saline in Postoperative Analgesia After Laparoscopic Hysterectomy: A Randomized, Double Blind, Placebo Controlled Trial
Brief Title: IV Acetaminophen for Postoperative Pain Analgesia After Laparoscopic Hysterectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Noah Rindos, Fellow in Minimally Invasive Gynecology, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PRO13110403
Record Dates: First submitted 2015-03-18; First posted 2015-03-27 (Estimated); Results first posted 2017-12-21 (Actual); Last update posted 2018-06-13 (Actual); Status verified 2018-05

CONDITIONS: Pain
Keywords: Laparoscopic Hysterectomy; IV acetaminophen; Postoperative pain control; Surgery
MeSH Terms: conditions — Pain | interventions — Acetaminophen; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intravenous IV acetaminophen (Experimental): The patients in the treatment arm will receive 1000mg of IV acetaminophen.
  Interventions: Drug: IV acetaminophen
- Normal Saline (Placebo Comparator): The patients in the placebo arm will receive normal saline.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: IV acetaminophen — The patients in the treatment arm will receive 1000mg of IV acetaminophen.
  Other Names: OFIRMEV
  Arms: Intravenous IV acetaminophen
Drug: placebo — The patients in the placebo arm will receive normal saline.
  Other Names: Normal saline
  Arms: Normal Saline

SUMMARY:
The objective of this study is to quantify the change in post-operative pain scores and narcotic requirements in women receiving pre and post-operative IV acetaminophen compared to placebo in women undergoing laparoscopic hysterectomy.

DETAILED DESCRIPTION:
Gynecologic surgery has been revolutionized by the incorporation of minimally invasive techniques. Procedures that once resulted in multiple day hospital admissions are now being performed in outpatient surgery centers. Common factors that contribute to delayed discharge are inadequate postoperative pain control and increased nausea and vomiting. A multi-modal pain management approach is considered optimal at controlling postsurgical pain, which includes combining different analgesics that act in varying mechanisms. By using medications that act synergistically, the overall analgesia requirement can oftentimes be decreased.

Opioids have been found to be highly effective in controlling postoperative pain; however, are associated with dose-dependent risks including nausea, vomiting, constipation, urinary retention, sedation, and respiratory depression. Subsequently, non-opioid options are frequently desired in an attempt to minimize narcotic intake. In the United States, intravenous acetaminophen was approved by the US Food and Drug Administration (FDA) in November 2010 for the management of mild to moderate pain and the reduction of fever. Since this time, multiple studies have analyzed the role of intravenous acetaminophen in both acute and postoperative pain; however, none have been specific to laparoscopic hysterectomy. The primary study published evaluating intravenous acetaminophen in laparoscopic hysterectomies also included multiple other laparoscopic procedures from a variety of specialties including general surgery, urology, and urogynecology. In addition, the intravenous acetaminophen was started on average 19 hours after the conclusion of the case once the patient controlled analgesic was discontinued.

Improved postsurgical pain control achieved with intravenous acetaminophen may potentially lead to same day discharge after major laparoscopic gynecologic procedures. Same day discharge after laparoscopic hysterectomy has been shown to be a safe option with proper patient counseling and multi-modal pain medications. In addition, same day discharge is also associated with decreased health care expenditures. With continued efforts to cut hospital costs, the pressure to discharge patients earlier continues to be high.

The investigators propose that intravenous acetaminophen will improve post-operative pain control and decrease narcotic requirements for patients undergoing laparoscopic hysterectomies. Furthermore, The investigators expect to find decreased postsurgical nausea and vomiting and potentially quicker discharge to home. This could have a large impact on the field of gynecologic surgery as major procedures that once required overnight admission may now succeed at same day discharge.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-75
* Ability to read and write in English (our post-operative pain log is only available in English)
* Planning a laparoscopic hysterectomy (includes total laparoscopic hysterectomy, laparoscopic supracervical hysterectomy, laparoscopically assisted vaginal hysterectomy, with or without salpingooophorectomy)

Exclusion Criteria:

* Answering yes to any of the following questions: "Do you have a history of liver disease, kidney disease, hepatitis C, history of liver failure, greater than 3 drinks per day or being have you ever been told by your doctor that they should not take acetaminophen"
* History of cardiac arrhythmia
* History of jaundice
* Acute abdominal inflammatory or infectious process at time of surgery
* Known malignancy at time of surgery
* Known pregnancy at time of surgery
* Plan to perform additional significant surgical procedure at the time of hysterectomy such as extensive excision of endometriosis on bowel or bladder or pelvic reconstructive procedure
* >6cm abdominal incision in order to remove the uterus at time of study-related hysterectomy
* Regular use of narcotic pain medication (defined as use on most days of the week at any point in the past 3 months)
* Allergy to acetaminophen
* Women who weigh less than 50 kilograms on the day of surgery.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2015-02; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Noah Rindos, MD, Principal Investigator — Faculty
Locations (1):
- Magee Womens Hospital, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Gonzalez AM, Romero RJ, Ojeda-Vaz MM, Rabaza JR. Intravenous acetaminophen in bariatric surgery: effects on opioid requirements. J Surg Res. 2015 May 1;195(1):99-104. doi: 10.1016/j.jss.2015.01.004. Epub 2015 Jan 14. PMID 25680474

RESULTS

PARTICIPANT FLOW:
Groups:
- Intravenous IV Acetaminophen: The patients in the treatment arm will receive 1000mg of IV acetaminophen.
  IV acetaminophen
- Normal Saline: The patients in the placebo arm will receive normal saline.
  placebo
Period: Overall Study
Arm/Group | Intravenous IV Acetaminophen | Normal Saline
Started | 91 | 92
Completed | 89 | 91
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intravenous IV Acetaminophen | Normal Saline | Total
Number analyzed (Participants) | 91 | 92 | 183
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 91 | 92 | 183
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91 | 92 | 183
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 91 | 92 | 183

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Pain
Description: The primary aim of this study is to compare overall post-surgical pain after hysterectomy as reported by the patients on a visual analog scale with a range of 0 to 10 where 0 is no pain at all and 10 is the worst pain that a person can imagine. Less pain is considered preferable to more pain. The theory is that patients who have intravenous acetaminophen will report less post-surgical pain.
Time Frame: 24 hours
Measure: Mean (95% Confidence Interval); unit: units on a visual analog scale
Arm/Group | Intravenous IV Acetaminophen | Normal Saline
Number analyzed (Participants) | 91 | 92
units on a visual analog scale | 3.55 [1.08 to 6.02] | 3.11 [0.89 to 5.33]

2. Secondary Outcome: Narcotic Medication Use
Description: The secondary outcome is comparison of narcotic pain medical requirements within the first 24 hours after surgery. The hypothesis is that the intravenous acetaminophen group will require less narcotic medications than the placebo group. Narcotic use in this study will be calculated by converting all narcotics (fentanyl, dilaudid etc) into standardized units of morphine using well validated conversion tables.
Time Frame: 24 hours
Population: This analysis is of the total number of units of morphine used by each group over a 24 hour period that is composed of the amount of narcotics received in the operating room, recovery room as well as at 6,12, and 24 hours postoperatively.
Measure: Mean (95% Confidence Interval); unit: Morphine Equivalents
Arm/Group | Intravenous IV Acetaminophen | Normal Saline
Number analyzed (Participants) | 89 | 91
Morphine Equivalents | 16.4 [4.9 to 27.9] | 18.4 [6.6 to 30.2]

3. Other Pre Specified Outcome: Having a Feeling of General Well-being at One Month
Description: Quality of recovery will be evaluated through the use of the validated Quality of Recovery-40 questionnaire. The hypothesis is that the intravenous acetaminophen group will experience an increased quality of recovery as compared to the placebo group.
Time Frame: 4 weeks
Population: The patients were asked to report their overall feeling of well being on a Visual Analog Scale one month after surgery. The scale has a range from 0 to 10 where a score of 0 would indicate the lowest (best) possible level of an outcome (pain, nausea etc) and a 10 would indicate the highest (worst) possible level.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Intravenous IV Acetaminophen | Normal Saline
Number analyzed (Participants) | 89 | 91
units on a scale | 4.11 [3.13 to 5.09] | 4.31 [3.37 to 5.25]

4. Other Pre Specified Outcome: Number of Participants Who Vomited Within 24 Hours of Operation
Description: A secondary aim of this study is to compare post-operative vomiting scores on post-operative day zero and one. Vomiting is reported as either having vomited or not vomited. The hypothesis is that the intravenous acetaminophen group will experience decreased vomiting compared with the placebo group.
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous IV Acetaminophen | Normal Saline
Number analyzed (Participants) | 91 | 92
Participants | 1 | 2
Statistical Analysis 1: Comparison: Intravenous IV Acetaminophen vs Normal Saline; Test type: Other; p = 0.517, Fisher Exact

5. Other Pre Specified Outcome: Readiness for Discharge
Description: Patient perception of satisfaction at time of discharge on post-operative day zero will be evaluated. The hypothesis is that intravenous acetaminophen group will experience increased satisfaction for discharge than the placebo group.
Time Frame: 24 hours
Population: Patients who were asked about overall satisfaction with procedure at time of discharge using a Visual Analog Scale. The scale has a range from 0 to 10 where a score of 0 would indicate the lowest (best) possible level of an outcome (pain, nausea etc) and a 10 would indicate the highest (worst) possible level.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Intravenous IV Acetaminophen | Normal Saline
Number analyzed (Participants) | 89 | 91
units on a scale | 7.76 [5.44 to 9.98] | 8.15 [5.97 to 10.33]

6. Other Pre Specified Outcome: Nausea Before Surgery as Compared to After Surgery
Description: A secondary aim of this study is to compare post-operative nausea on post-operative day zero and one as reported by the patients on a visual analog scale with a range of 0 to 10 where 0 is no nausea at all and 10 is the worst nausea that a person can imagine. Less nausea is considered preferable to more nausea. The hypothesis is that the intravenous acetaminophen group will experience decreased nausea compared with the placebo group.
Time Frame: 24 hours
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Intravenous IV Acetaminophen | Normal Saline
Number analyzed (Participants) | 91 | 92
units on a scale | 0.69 [-0.56 to 1.94] | 0.85 [-0.73 to 2.43]
Statistical Analysis 1: Comparison: Intravenous IV Acetaminophen vs Normal Saline; Test type: Other; p = 0.508, Fisher Exact

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | Intravenous IV Acetaminophen | Normal Saline
All-Cause Mortality (participants affected / at risk) | 0/91 | 0/92
Serious Adverse Events (participants affected / at risk) | 1/91 | 0/92
Other Adverse Events (participants affected / at risk) | 10/91 | 11/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intravenous IV Acetaminophen (N=91) | Normal Saline (N=92)
In patient hospitalization (Vascular disorders) | 1 (1) | 0 (0) — Postoperatively there was concern that the patient had undergone a cerebrovascular accident (CVA). She was withdrawn from the study and admitted to the intensive care unit. An extensive workup was performed with no evidence of any adverse event.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intravenous IV Acetaminophen (N=91) | Normal Saline (N=92)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2) — Patients who reported episode of vomiting at 24 hours
Pain (Nervous system disorders) | 1 (1) | 0 (0) — The patient had postoperative pain, withdrew from the study. The second dose of study medication was not given.
Nausea (Gastrointestinal disorders) | 8 (8) | 9 (9) — Reports of nausea with level greater than 2 out of 10 at 24 hours.

LIMITATIONS AND CAVEATS:
The original protocol involved 154 patients with an expected rate of loss to follow up of 10%. Due to higher than expected loss to follow up the number of patients enrolled was increased to 190.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes